CLINICAL TRIAL: NCT00733447
Title: SynCardia Freedom Driver System Study
Status: Approved for marketing | Type: Expanded Access
Sponsor: SynCardia Systems. LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: RA-142; P030011
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Biventricular Failure
Keywords: Biventricular failure
MeSH Terms: interventions — Drug Delivery Systems

INTERVENTIONS:
Device: CardioWest temporary Total Artificial Heart (TAH-t) System — The SynCardia CardioWest temporary Total Artificial Heart (TAH-t) System is a pulsatile biventricular device that replaces a patient's native ventricles and valves, and pumps blood to both pulmonary and systemic circulation. The system consists of the implantable CardioWest TAH-t and an external pneumatic driver connected by drivelines.

SUMMARY:
The purposes of this study are to confirm that the Freedom Driver System is a suitable pneumatic driver for clinically stable TAH-t subjects, and that patients and lay caregivers can be trained to manage the Freedom Driver System safely outside the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are implanted with the TAH-t and are clinically stable.

Exclusion Criteria:

* Patients who are implanted with the TAH-t and are not clinically stable.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2010-03; Primary Completion 2013-08 (Actual); Study Completion 2014-05 (Estimated)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Virginia Commonwealth University Medical Center, Richmond, Virginia